CLINICAL TRIAL: NCT00855296
Title: Thrombin Regulated Platelet Activation
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Heidi Hamm, Professor and Chair of Pharmacology, Vanderbilt University
Other Study IDs: 050182
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Thrombin is the most potent activator of platelets, and platelet activation is a hallmark of thrombosis. Coronary artery disease (CAD) is the major cause of mortality and morbidity in the United States and other industrialized countries, and thrombotic sequelae are the key cause of death in diabetes. The accumulation of thrombin at sites of vascular injury provides one of the major mechanisms of recruiting platelets into a hemostatic plug. Thrombin works by activation of the G protein-coupled protease activated receptors PAR1 and PAR4 on human platelets to initiate signaling cascades leading to increases in [Ca]i, secretion of autocrine activators, trafficking of adhesion molecules to the plasma membrane, and shape change, which all promote platelet aggregation. The thrombin receptors work in a progressive manner, with PAR1 activated at low thrombin concentrations, and PAR4 recruited at higher thrombin concentrations. As direct thrombin inhibitors become widely used in clinical practice, it is important to assess their effects on vascular function. Our hypothesis is that PAR1 and PAR4 do not signal through the same G protein pathways, and that PAR4 is not a strong platelet agonist. To investigate this hypothesis, the investigators will study the G protein pathways downstream of PAR4, and assess ex-vivo platelet responsiveness to thrombin, PAR1, and PAR4 agonist peptides, both in normal human subjects, and along the stages of pathology, from patients with stable angina as well as unstable angina who are undergoing angioplasty. Similarly, the investigators will examine platelet function in patients with metabolic syndrome as well as diabetes, along the continuum from insulin resistance to full-blown disease. These studies will provide deeper insight into the G protein pathways used by PARs. They will elucidate the contribution of PAR receptors to normal platelet function as well as the abnormal platelet activation in thrombotic states. The long term goal is to understand the implications for PAR receptors as therapeutic targets for anti-platelet therapies that may carry less bleeding risk.

DETAILED DESCRIPTION:
Thrombin is the major protease in the coagulation cascade whose pleiotropic actions can ultimately lead to thrombosis and tissue injury. Thrombin is the key effector of the coagulation cascade and converts fibrinogen to fibrin which is essential for laying the mesh work for clot formation. Further, thrombin also provides positive feedback by converting inactive coagulation factors into their active state, thereby generating more thrombin. In addition, thrombin displays a diverse range of effects in vascular cells that functionally connects tissue damage to both hemostatic and inflammatory responses. Many of the cellular effects of thrombin are initiated via activation of a family of Protease-Activated Receptors (PARs) which are coupled to heterotrimeric G proteins.

Cardiovascular disease remains the leading cause of death in the United States, accounting for over 39% of deaths and over $350 billion in annual health care costs in this country. Current pharmacological therapy for treatment of diseases caused by blood clots, such as heart disease and stroke, often involve the use of drugs that do not reflect current scientific understanding of these pathologies. Acute coronary syndrome is a thrombotic event, and platelet activation plays a critical role in the formation of intravascular thrombus at the site of arterial injury or plaque rupture. Medical management of acute coronary syndrome is centered on anti-platelet therapies, however, current anti-platelet drugs do not fully attenuate platelet activation, can have delayed onset and long durations of action and may result in significant morbidity due to bleeding complications. With increasing numbers of percutaneous coronary intervention in patients with ACS, bleeding complications become a major concern in this new era of anti-platelet and coagulation therapies. The direct thrombin inhibitor bivalirudin was associated with a significant reduction of in-hospital bleeding complication as compared to heparin plus IIbIIIa inhibitors in patients undergoing PCI, while composite clinical endpoints (death, MI, repeated revascularization) were maintained. An explanation for the lack of superiority of direct thrombin inhibitors when compared to heparin, could be that direct thrombin inhibitors also block the anticoagulation and anti-inflammatory effects of thrombin thereby potentially altering the risk/benefit ratio. In addition, all of the agents used in treating ACS have undesirable side effects such as bleeding. An agent that would selectively block the inflammatory and thrombotic effects of thrombin by selectively blocking PAR activation, without altering the protective APC pathway or inhibiting fibrin generation (bleeding) would potentially have more of a desirable risk/benefit ratio.

Given the known roles of proteases and PARs in coagulation, inflammation, pain, healing and protection, the need for development of a PAR antagonist as a therapeutic agent for treatment of thrombosis, atherosclerosis and inflammation is well-recognized. Thus, blocking PAR action by inhibiting the PAR-G protein interface is an alternative target for blocking downstream consequences of thrombin-mediated cellular activation. Since there are two PARs on human platelets, PAR1 and PAR4, it is critical to define the roles of both receptors in several likely clinical settings where PAR antagonists would be used. In this proposal both the G protein pathways underlying PAR signaling mechanisms as well as their roles in pathologies characterized by activated platelets will be studied in detail. We propose in this grant to investigate the specific roles of individual PARs in mediating the events leading to the multi-stage process of platelet activation and clot formation. The long term goals of these studies are to determine novel PAR-specific anti-platelet therapies.

In defining which G protein mediates the effects of different PARs on platelets, we will target that particular receptor-G protein interface using the C-terminus of the particular G alpha that mediates the response. We have used overexpression of the native C-terminal peptides of different G proteins to determine which G protein signaling pathway is involved in physiological responses in endothelial cells. As this method is not applicable to platelets, which are not transfectable, we propose to create membrane-permeable versions of Gα C-terminal peptides that would be acutely deliverable to platelets to tease out signaling pathways. The roles of G proteins in platelet activation in mice has been studied extensively through the use of knockout technology. The most striking phenotype was in mice lacking G alpha q. They demonstrate an absence of platelet aggregation and are protected against thromboembolism. Recently, the role of G alpha 13 in platelets has been uncovered through the use of an inducible mouse line lacking G alpha 13. Previously the role of G alpha 13 was unknown as these mice die in utero from defects in angiogenesis. Surprisingly, absence of G13 in mice platelets leads to a reduced potency of thrombin, TXA2 and collagen to induce platelet shape change and aggregation. The specific roles of G proteins in platelet activation in humans has been less well studied, because of the lack of a tractable genetic approach and the inability to transfect human platelets. One study has identified a patient with diminished Gαq activity (50% of Gαq immunoreactivity compared to normal) who also had impaired agonist-induced platelet aggregation and secretion.

Significant differences exist in the expression patterns of G proteins and PARs between mouse and human platelets. Perhaps the biggest difference is that thrombin activation of mouse platelets is mediated through PAR3 and PAR4, while thrombin activation of human platelets is mediated through PAR1 and PAR4. This was made very clear as thrombin was still able to activate platelets in PAR1 knockout mice. Murine PAR3 is unable to signal to downstream effectors and functions to present thrombin to PAR4 in platelets, as PAR4 lacks the hirudin-like sequence and does not bind thrombin efficiently. By contrast, human PAR3 has been proposed to signal through thrombin-triggered phosphoinositide hydrolysis, however, its functional role remains to be established. Mice platelets only express Gαq while not expressing Gα11, which most likely explains the more severe phenotype with Gαq knockout mice compared to the other knockout mice. However, human platelets may contain G alpha 11, in addition to G alpha q, although this has been viewed with controversy. Our dominant-negative G protein peptide strategy should now allow us to directly study PAR-G protein signaling in human platelets.

Coronary artery disease (CAD) is the leading cause of death in the world. The lifetime risk of having coronary heart disease after age 40 is 49% for men and 32% for women. The AHA estimates that more than 12 million people have some form of CAD history. This will increase with the aging of the baby boom generation. Research spanning nearly three decades has firmly established the role of platelet activation in the pathophysiology of ACS. In contrast to the central role of platelet activation in the pathogenesis of unstable angina and acute myocardial infarction, a major role for platelet activation in the setting of chronic stable angina has not been widely acknowledged. Coronary angioplasty leads to vessel wall injury and exposure of subendothelial structures with resultant platelet activation that may limit the early and late success of the procedure. In contrast with the findings in patients with stable angina, patients referred for angioplasty exhibit more consistent increases in platelet activation prior to their intervention. Platelet aggregation and the expression of activated GPIIbIIIa and P-selectin are increased in patients referred for coronary artery stenting or angioplasty. In contrast, increased concentrations of circulating markers of platelet activation in patients following angioplasty have been reported by some but not all groups. Based on the REPLACE-2 trial of bivalirudin, interventional cardiologists at Vanderbilt and around the world are increasingly using bivalirudin as the anticoagulant of choice for PCI. We will examine the effects of blocking thrombin on PAR signaling in platelets from subjects with normal coronary arteries as well as patients undergoing PCI. We have carried out preliminary studies of platelet aggregation before and after bivalirudin infusion in patients from Vanderbilt's Coronary Catheterization Laboratory. As expected, thrombin mediated aggregation of ex vivo platelets is inhibited by bivalirudin (data not shown). Therefore, we hypothesize that removing the protective effect of basal thrombin on the vasculature could change the platelet PAR1 or PAR4 signaling state. This possibility has not been examined, and it is important that such studies be conducted, as direct thrombin inhibition becomes a more widely used therapeutic strategy in acute coronary syndrome.

These studies were designed to study PAR signaling and G protein activation states in patients with platelet activation in the setting of the continuum of the metabolic syndrome and diabetes mellitus. The degree of platelet activation as determined by assays of platelet reactivity and by the expression of markers of platelet activation will be correlated with the changes in PAR signaling. These studies will provide a comprehensive assessment of platelet activation in the setting of the metabolic syndrome, and will compare the extent of activation in this setting with that in a group of contemporaneously studied patients with diabetes mellitus. Finally, the influence of the direct thrombin inhibitor, bivalirudin on platelet activation and signaling will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18, Sex: male and female.
* Patients who undergo clinically indicated coronary angiography and/or PCI. Patients in Group 1 (elective PCI) include those presented with stable angina (ACC definition for stable angina).
* Coronary angiography reveals severe stenosis (>70%) that requires PCI.
* Patients in Group 2 (elective PCI in subjects with diabetes) include those who present with stable angina, or with findings on non-invasive testing (exercise or pharmacologic stimulation with imaging by nuclear perfusion imaging or stress echocardiography) in whom coronary angiography reveals severe stenosis (>70%) that requires PCI.
* Patients in Group 2 (ACS) include those presented with unstable angina or non-ST elevation myocardial infarction (as defined by the ACC).
* Coronary angiography reveals severe stenosis (>70%) that requires PCI.

Exclusion Criteria:

* Significant left main coronary artery disease.
* Severely impaired left ventricular systolic function (EF<35%).
* Prior treatment with enoxaparin, Bivalirudin (or other thrombin inhibitors), Warfarin, or thrombolytic agents <48 hours.
* Prior history of myocardial infarction (<6 weeks). Prior history of stroke (<6 weeks).
* Prior history of coronary intervention (<6 weeks).
* History of HIV/AIDS.
* The patients will be identified in the following manner:
* All subjects will be picked from a pool of patients diagnosed with stable angina and diabetes from the Vanderbilt Page-Campbell Heart Institute at Vanderbilt University Medical Center and undergo a complete history and physical examination.
* Patients with acute coronary syndrome will be referred from the acute cardiology patient service at Vanderbilt University Medical Center.
* Subjects with hematologic, renal (creatinine > 2.0 mg/dl), hepatic, inflammatory, and neoplastic disorders, and those who sustained a recent (< 1 month) myocardial infarction, ACS, or stroke will be excluded. Patients who used nonsteroidal anti-inflammatory drugs, corticosteroids, or hormone replacement therapy will also be excluded.
* Pregnancy will be excluded in women of child bearing potential by measurement of urine ß-HCG (it is standard of care to determine if a woman is pregnant prior to elective PCI and will be screened as part of their PHI).
* For healthy volunteers, pregnancy will be excluded per verbal report.
* Data will be collected regarding patient demographics including height and weight, abdominal circumference, blood pressure, comorbid medical conditions, triglycerides, HDL, fasting glucose and medication use (including prescription of antithrombotic agents, ACE inhibitors, angiotensin receptor blockers, beta blockers, calcium channel antagonists and HMG-CoA inhibitors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing angioplasty
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2006-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi E. Hamm, Ph.D., Principal Investigator — Vanderbilt Universtiy Medical Center, Pharmacology
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States